CLINICAL TRIAL: NCT06877000
Title: Vitiligo Severity, Quality of Life, Work Productivity and Activity Impairment Among Patients in Upper Egypt
Brief Title: Vitiligo Severity, Quality of Life, Work Productivity and Activity Impairment
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Salah Ahmed Abdelhady, Resident, Assiut University
Other Study IDs: Vitiligo quality of life
Record Dates: First submitted 2025-03-06; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Working vitiligo patient: Employed moderate to severe vitiligo patients
  Interventions: Other: VITIQOL questionnaire
- Working not diseased individuals: Employed healthy individuals

INTERVENTIONS:
Other: VITIQOL questionnaire — 16 questions questionnaire measure effect of vitiligo on quality of life
  Other Names: WPAI questionnaire and GSE scale
  Groups: Working vitiligo patient

SUMMARY:
translate and validate the vitiligo specific quality of life (VITIQOL) questionnaire to Arabic language.

evaluate the effect of vitiligo on patient quality of life using vitiligo specific quality of life questionnaire (VitiQoL).

measure the impact of vitiligo on work productivity using work productivity and activity impairment questionnaire (WPAI) and general self efficacy scale (GSE) .

analyze how disease severity and location influence patients quality of life and work pro

DETAILED DESCRIPTION:
Vitiligo is a common disorder of depigmentation caused by the progressive destruction of melanocytes that affect the skin, hair and mucous membranes, clinically presenting as depigmented macules and leukotrichia.

Vitiligo was historically regarded as a cosmetic disorder; however, it is an immune disease as it affects patient well-being . It affects approximately 0.5-1% of the global population. A Study reported a prevalence of 1.2% in the Egyptian population.

Vitiligo is asymptomatic disease, so its effect on quality of life is much more related to psychological problems, such as lack of self-confidence unpleasant body images unsuccessful social relationships, and lower quality of marital relations, than the exclusive physical issues. It has been shown that patients with vitiligo are at risk of higher social discrimination and stigma Lesions that are more severe, on the face, or covering a greater BSA are more often associated with poorer outcomes and activity impairment.

Recently a study conducted in Egypt in 2023 noted that more than half of studied sample had low level of self-esteem and quality of life. While more than half of studied sample had moderate negative body image. Also, half of studied sample had moderate level of social problems .

limited studies have been conducted in Upper Egypt which assess life quality of patients with vitiligo and but those Studies employed non-specific tools like Dermatology Life Quality Index (DLQI).

Lilly et al have developed a reliable tool with high internal consistency named as Vitiligo specific Quality of life questionnaire(VITIQOL) that consists of 16 questions comprising of demographic and clinical parameters of the patients.

Also the work productivity and activity impairment among vitiligo patients in Egypt have not been assessed before .

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years and less than 60 years old diagnosed with vitiligo by a physician Patients willing to complete the survey questionnaires Patients who can speak Arabic

Exclusion Criteria:

* Patients with other major skin disease affecting QOL . Patient with chronic diseases as diabetes mellitus and hypertension Not working patients

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: 200 cases and 200 control will be selected from vitiligo clinic Assiut university
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Arabic validated version of vitiligo specific quality of life instrument VITIQOL | Baseline
  A translated version will help to measure impact of vitiligo in Arabs
Patients with severe vitiligo which will be measured by vitiligo area scoring index VASI score , will have lower quality-of-life on vitiligo specific quality of life instrument which have a score ranges from 0 to 90 | Baseline
  Vitiligo specific quality of life instrument have 15 questions each one has a likert scale from 0 to 6 , score ranges from 0-90 , patients with severe vitligo expect to have low score on the questionnaire
patients with more severe vitiligo have low work productivity and more activity impairment | Baseline
  Work Productivity and Activity impairments questionnaire is a 6 question questionnaire consists of four consists of four metric :
  1. Absenteeism (the percentage of work time missed)
  2. Presentism (the percentage of impairment experienced while at work)
  3. Overall work productivity loss (an estimate of combination of absenteeism and presentism)
  4. Activity impairment (the percentage of impairment in daily activities) WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity .

CONTACTS AND LOCATIONS:
Overall Officials: Esraa Sa Ahmed, Resident, Principal Investigator — Assiut University

REFERENCES:
- [Background] Attallah, D. A., Abdullah, M. A. A., & Abou-Taleb, D. A. E. (2022). Effect of treatment on quality of life in Egyptian vitiligo patients using the Arabic version of Dermatology Life Quality Index. Journal of Current Medical Research and Practice, 7(2), 163-166.
- [Background] Lilly E, Lu PD, Borovicka JH, Victorson D, Kwasny MJ, West DP, Kundu RV. Development and validation of a vitiligo-specific quality-of-life instrument (VitiQoL). J Am Acad Dermatol. 2013 Jul;69(1):e11-8. doi: 10.1016/j.jaad.2012.01.038. Epub 2012 Feb 25. PMID 22365883
- [Background] Rosmarin D, Soliman AM, Piercy J, Marwaha S, Anderson P, Camp HS. Health-Related Quality of Life Burden Among Adults with Vitiligo: Relationship to Disease Severity and Disease Location. Dermatol Ther (Heidelb). 2024 Jun;14(6):1633-1647. doi: 10.1007/s13555-024-01187-z. Epub 2024 Jun 2. PMID 38824482